CLINICAL TRIAL: NCT07112274
Title: Effect of Empagliflozin on Cardiac Remodeling in Non Diabetic Patients With Preserved Heart Failure
Brief Title: Empagliflozin on Patients With Preserved Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMPAGLIFLOZIN on HF
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: All participants will be randomly divided into two groups: group (A) for empagliflozin (n=25), group (B) for placebo (n=25)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin Group (Experimental): group (A) for empagliflozin (n=25),
  Interventions: Drug: Empagliflozin 10 MG
- Placebo Group (Placebo Comparator): group (B) for placebo (n=25)
  Interventions: Other: Placebo Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Treatment group will receive empagliflozin 10 mg tablet once daily
  Other Names: Mellitofix
  Arms: Empagliflozin Group
Other: Placebo Tablet — control group will receive placebo tablet.
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
The proposed research in this application will investigate the effect of empagliflozin on cardiac remodeling in patients with heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. About 50 cardiac non diabetic patients diagnosed with heart failure with preserved ejection fraction will be recruited from Mahalla Cardiac Centre outpatient clinics and randomize them into two groups, group on empagliflozin 10 mg once daily and the second group placebo.
4. Blood samples will be collected before, and 3 months after intiation of the trial for evaluating Complete blood count (CBC), Serum creatinine (SCr), Aspartate aminotransferase (AST), Alanine transaminase(ALT), Hemoglobin A1C and two biomarkers which are: Human N-Terminal Pro Brain Natriuretic Peptide (NT-ProBNP) and soluble suppressor of tumorigenicity 2 (sST2) values in both groups.
5. Echocardiogram will be assessed for the patients before and 3 months after the initiation of study and the values of :

   1. Left ventricular end systolic volume index (LVESI)
   2. Left atrial volume index (LAVI)
   3. Left ventricular mass index (LVMI)
   4. Ejection fraction (EF)
   5. Left atrium size
   6. Grade of diastolic dysfunction
   7. Cardiac output (C.O.P)
   8. Stroke volume (SV)

      Method:

      - All participants will be randomly divided into two groups: group (A) for empagliflozin (n=25), group (B) for placebo (n=25)

      Sample sizes of 50 cardiac patients (25 empagliflozin group and 25 placebo group), achieves 90% power to detect a difference (7.5 ml/m2) in the mean change of Left ventricular end systolic volume index (LVESI) between the 2 groups, using independent t test, at a 0.05 significance level.

      The sample size was calculated using NCSS 2004 and PASS 2000 software
      * Treatment group will receive empagliflozin 10 mg tablet once daily and control group will receive placebo tablet.
      * Cardiac biomarkers will be assessed at baseline before trial initiation and 3 months after the initiation of trial
      * SPSS will be used for statistical analysis of the data obtained in the research, measurement data using t test
      * A value of P<0.05 was considered to indicate a statistically significant difference.

ELIGIBILITY:
Inculsion

1. Cardiac patients who diagnosed with HFpEF, EF more than 50 %.
2. Patients should have basically normal liver and kidney functions, normal coagulation, and have no serious auditory, visual or central nervous system diseases.
3. Patients with no history of immune system disease.

Exclusion

1. Patients with declined baseline creatinine clearance below 60 ml/min
2. Patients diagnosed with acute liver failure, AKI, hypoglycemia.
3. Allergy to the ingredients which will be used in this study
4. Patients with Diabetic ketoacidosis or non ketotic hyperosmolar hyperglycemia
5. Severe hepatic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
NT-ProBNP | 3 months
  Human N-Terminal Pro Brain Natriuretic Peptide (NT-ProBNP)
sST2 | 3 months
  soluble suppressor of tumorigenicity 2 (sST2)

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malik A, Brito D, Vaqar S, et al. Congestive Heart Failure. [Updated 2022 May 5]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2022 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK430873/
- [Background] Lee MMY, Brooksbank KJM, Wetherall K, Mangion K, Roditi G, Campbell RT, Berry C, Chong V, Coyle L, Docherty KF, Dreisbach JG, Labinjoh C, Lang NN, Lennie V, McConnachie A, Murphy CL, Petrie CJ, Petrie JR, Speirits IA, Sourbron S, Welsh P, Woodward R, Radjenovic A, Mark PB, McMurray JJV, Jhund PS, Petrie MC, Sattar N. Effect of Empagliflozin on Left Ventricular Volumes in Patients With Type 2 Diabetes, or Prediabetes, and Heart Failure With Reduced Ejection Fraction (SUGAR-DM-HF). Circulation. 2021 Feb 9;143(6):516-525. doi: 10.1161/CIRCULATIONAHA.120.052186. Epub 2020 Nov 13. PMID 33186500